CLINICAL TRIAL: NCT06347263
Title: Clinical and Radiographic Evaluation of Using the Entire Papilla Preservation Technique With and Without Autogenous Bone Graft and Injectable Platelet Rich Fibrin in Treatment of Periodontal Intraosseous Defects: A Randomized Clinical Tria
Brief Title: Clinical and Radiographic Evaluation of Using the Entire Papilla Preservation Technique With and Without Autogenous Bone Graft and Injectable Platelet Rich Fibrin in Treatment of Periodontal Intraosseous Defects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Laila Taher Sedeek Mohamed, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PER 332
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Isolated Intrabony Periodontal Defects in Patients With Periodontitis
Keywords: Periodontal intrabony defects; Entire papilla preservation technique; EPPT; Injectable platelet rich fibrin; I-PRF

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding of the operator and patient is not applicable.
  - Outcome assessor (primary and secondary outcomes) & biostatistician will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Procedure:Entire papilla preservation technique with autogenous bone and injectable platelet rich fibrin
  Interventions: Other: Entire papilla preservation technique
- Control group (Active Comparator): Procedure: Entire papilla preservation technique alone.
  Interventions: Other: Entire papilla preservation technique

INTERVENTIONS:
Other: Entire papilla preservation technique — Minimally invasive periodontal surgery

SUMMARY:
The goal of this Clinical trial is to evaluate the clinical and radiographic outcomes of using entire papilla preservation technique with and without autogenous bone and injectable platelet rich fibrin in treatment of isolated Intrabony defects in patients with stage III periodontitis.

DETAILED DESCRIPTION:
Research objective: The aim of conducting this research is the development of a newer, less invasive and cost-effective surgical approaches that help in treatment of periodontal intrabony defects.Due to the shortcomings of access flap approaches , another minimally invasive surgical technique which is the Entire papilla preservation technique will be used to approach the defect .Also, due to the short comings of using other bone substitute materials and resorbable membranes , the Autogenous bone graft which is the gold standard of bone grafts and the injectable platelet rich fibrin will be used in this study .

Research Procedure in brief:

The study is to be conducted in the Oral Medicine and Periodontology department, Faculty of Dentistry - Cairo University, Egypt. This study will be carried out on patients enrolled from the Outpatient Clinic of Oral Medicine and Periodontology department, Faculty of Dentistry, Cairo University.

Eligibility criteria:

I. Inclusion criteria:

1. Patients with healthy systemic condition.
2. Adult patients (18 years old and older).
3. Patients with stage lll periodontitis, having one isolated intrabony defect with probing depth >6 mm, clinical attachment level> 6 mm and at least 4 mm intrabony component involving predominantly the interproximal area of the affected tooth.
4. Patients with full mouth plaque score<20%.
5. Patients with full mouth bleeding score<20%.
6. Compliance with good oral hygiene.
7. Patients accept 6-months follow-up period (cooperative patients).
8. Patients provide an informed consent.

II. Exclusion criteria:

1. Ongoing drug therapy that might have an impact on the clinical signs and symptoms of periodontitis.
2. One wall intrabony defect.
3. Defects that involve the buccal and lingual sites.
4. Smokers ˃ 10 cigarettes / day.
5. Pregnant and lactating females.

General operative procedures:

1.Preoperative preparation:

Clinical examination:

Each patient will be examined to confirm that he/she met the eligibility criteria. This is followed by:

1. Full mouth charting to evaluate the periodontal status will be performed by using UNC 15 periodontal probe, including assessment of plaque index (PI), bleeding on probing (BOP), probing depth (PD), clinical attachment level (CAL), gingival recession, and radiographic x-ray imaging.
2. Patients will be thoroughly informed on self-performed plaque control activities consisting of using the modified Bass brushing technique, a soft toothbrush, regular toothpaste twice a day, and inter-dental cleaning once a day.
3. The patients will receive supra gingival scaling with ultrasonic scaler, then they will be recalled after 2 weeks. 4_An oral hygiene session will be performed two weeks before the surgical treatments.

Each patient will be prescribed a 0.2% chlorhexidine-based mouthwash, twice a day, for two weeks. Clinical photographs: Clinical photographs will be taken at baseline and at 12 months postoperatively. Radiographic examination: Periapical radiographs using paralleling technique using KCP film holder will be performed for each patient on the defect site to evaluate alveolar bone loss using DIGORA system.

Initial Therapy:

The initial therapy will consist of periodontal treatment (phase I therapy) including supra gingival scaling, subgingival debridement if needed, adjustment of faulty restoration and polishing. The mechanical plaque control instructions for each patient include brushing and interdental cleaning techniques.

Re-evaluation phase:

* 4-6 weeks after the initial therapy, periodontal re-evaluation will be done to confirm the sites that will require surgical therapy.
* Criteria used to indicate that surgery is required include the persistence of interproximal defect with PD ≥ 5 mm, CAL ≥ 4 mm.
* An individually customized positioning stent will be fabricated for each patient and a pre-operative periapical x-ray using parallel-angle technique will be employed using X-ray film holding system to ensure accuracy and reproducibility of the measurements.

Surgical procedures

* Pre-procedural mouth rinse using 0.2% chlorhexidine gluconate3 rinses for intraoral antisepsis.
* Surgical sites will be anaesthetized using local anesthesia.
* Following a buccal intra-crevicular incision, a bevelled vertical releasing incision will be performed in the buccal gingiva of the neighbouring inter-dental space and extended just beyond the mucogingival line( The Entire papilla preservation technique_EPPT)to provide adequate mechanical access to the intra-bony defect. A microsurgical periosteal elevator will be used to elevate a buccal full-thickness mucoperiosteal flap extending from the vertical incision to the defect-associated papilla.
* The inter-dental papilla will be elevated in full-thickness manner up to the intact lingual bone crest.
* A microsurgical scissor and mini curettes will be used to remove the granulation tissue from the inner aspect of the defect-associated inter-dental papilla.
* Any residual subgingival plaque or calculus will be gently removed from the exposed root surface with an ultrasonic scaler.
* The surgical site will be thoroughly rinsed with sterile saline.

The participants will be divided into two groups:

Intervention group:

* The Entire papilla preservation surgical technique (EPPT) will be performed to approach the intra-bony defects, with autogenous bone graft mixed with injectable platelet rich fibrin (I-PRF) placement. The graft will be harvested from the retromolar area using automatic chip maker (ACM) bur and a hand bone mill will be used to grind the chips into particles, then it will be mixed with I-PRF and placed in the defect.
* I-PRF will be prepared as follows:(Choukroun et al., 2018) 10 ml of peripheral venous blood will be collected into a sterile 10 ml plastic PRF tube (to reduce clotting time) without anticoagulants and centrifuged immediately at room temperature using centrifugal force 700 rpm for 3 minutes (60gRCF), then the yellow fluid (liquid fibrinogen) at the top of the tubes will be aspirated with a blunt sterile syringe, avoiding red blood cells.

Control group:

* The Entire papilla preservation surgical technique (EPPT) will be performed to approach the intra-bony defects without autogenous bone graft and Injectable platelet rich fibrin placement.
* For both groups, flaps will be approximated and sutured at the original position with a 5-0 or 6_0 monofilament polypropylene suture material. Postoperative Care
* Participants will be given instructions to avoid any trauma to the surgical site, refrain from interfering with the sutures, and to avoid consuming hot food or engaging in vigorous rinsing.
* They will be advised to continue tooth brushing for the other parts of their dentition, while gentle tooth brushing for the surgical site will be advised to be resumed after a two-week period.
* The patients will be requested to rinse gently with 0.12% chlorhexidine digluconate mouth rinse for 1 minute twice daily for a duration of two weeks.
* Participants will be prescribed either Amoxicillin 500 mg (Misr Co. for Pharmaceutical Industries, Egypt) three times daily for five days, or doxycycline 100mg (Doxycycline, Nile Co. for Pharmaceuticals and Chemical Industries, Egypt) twice daily if they have allergy to penicillin.
* Sutures will be removed two weeks after the surgery.
* All the subjects will be evaluated at 1, 3, 6 and 12 months for clinical and radiographic parameters. Outcomes:The results of Clinical attachmentlevel (CAL) gain, Linear bone fill, Gingival index (GI), Plaque index (PI), Probing pocket depth (PPD), Gingival recession (GR), Bleeding on probing (BoP), Postoperative pain and Patient satisfaction will be measured at baseline, 1 month, 3 months, 6 months and after 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with healthy systemic condition.
2. Adult patients (18 years old and older).
3. Patients with stage lll periodontitis, having one isolated intrabony defect with probing depth >6mm, clinical attachment level> 6mm and at least 4 mm intrabony component involving predominantly the interproximal area of the affected tooth.
4. Patients with full mouth plaque score<20%.
5. Patients with full mouth bleeding score<20%.
6. Compliance with good oral hygiene.
7. Patients accept 6-months follow-up period (cooperative patients).
8. Patients provide an informed consent.

Exclusion Criteria:

1. Ongoing drug therapy that might have an impact on the clinical signs and symptoms of periodontitis.
2. One wall intrabony defect.
3. Defects that involve the buccal and lingual sites.
4. Smokers ˃ 10 cigarettes / day.
5. Pregnant and lactating females.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level (CAL) gain change from baseline to 12 months | CAL gain will be taken at baseline, 3 month, 6 months and 12 months after the intervention during the follow-up period and will be done by a single calibrated examiner.]
  The CAL will be clinically measured using UNC 15 periodontal probe from the cemento-enamel junction (CEJ) to the depth of defect. An individually customized positioning stent will be fabricated for each patient to ensure accuracy and reproducibility of the measurements.

SECONDARY OUTCOMES:
Linear bone fill change from baseline to 12 months | Linear bone fill will be measured at baseline, 6 months and 12 months after the intervention during the follow-up period and will be done by a single calibrated examiner]
  Linear bone fill will be radiographically measured from the CEJ to the deepest part of the intrabony defect using the linear measurement tool of the Digora software. Individually customized positioning stent will be fabricated for each patient and parallel-angle technique will be employed using X-ray film holding system. This will ensure accuracy and reproducibility of the measurements. Radiographic linear defect depth (RLDD) will be measured as the depth of the intrabony defect from the alveolar crest to the defect base at baseline and 6 months postoperatively. The defect angle will be measured at baseline, as the angle formed between intersections of lines from the alveolar crest to the defect base and tooth long axis line. Calculation of bone fill in mm will be done by a subtraction of follow-up from baseline RLDD values, and percentages of bone fill will be expressed as the proportion of change to baseline RLDD.

CONTACTS AND LOCATIONS:
Overall Officials: Laila T Sedeek, Bachelor, Principal Investigator — Cairo University; Manal M Hosny, Professor, Study Director — Cairo University
Locations (1):
- Faculty of dentistry, Cairo University, Cairo, Egypt